CLINICAL TRIAL: NCT01394783
Title: Videolaryngoscope vs Classic Laryngoscope in Teaching Neonatal Endotracheal Intubation: a Randomized Controlled Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Moussa, Dr Ahmed Moussa, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 3282-CER
Record Dates: First submitted 2011-05-31; First posted 2011-07-14 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Intubation, Intratracheal
Keywords: Endotracheal intubation, Teaching, Videolaryngoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Classic laryngoscope (Other): Phase 1 and 2: Endotracheal intubation using the classic laryngoscope with Miller blade 0 or 1 according to weight of infant.
  Interventions: Device: Miller laryngoscope
- Videolaryngoscope (Other): Phase 1: Endotracheal intubation using the videolaryngoscope with blade 0 or 1 according to weight of infant. videolaryngoscope will be used to proceed to endotracheal intubation indirectly with the use of the video monitor for guidance. Phase 2: Endotracheal intubation using the classic laryngoscope with Miller blade 0 or 1 according to weight of infant.
  Interventions: Device: Storz videolaryngoscope

INTERVENTIONS:
Device: Miller laryngoscope — Phase 1 and 2: Endotracheal intubation using the Miller laryngoscope with blade 0 or 1 according to weight of infant.
  Arms: Classic laryngoscope
Device: Storz videolaryngoscope — Phase 1: Endotracheal intubation using the videolaryngoscope with blade 0 or 1 according to weight of infant. Videolaryngoscope will be used to proceed to endotracheal intubation indirectly with the use of the video monitor for guidance. Phase 2: Endotracheal intubation using the classic laryngoscope with Miller blade 0 or 1 according to weight of infant.
  Arms: Videolaryngoscope

SUMMARY:
Every year thousands of neonates born in North America need extensive resuscitation which often includes endotracheal intubation (ETI). In these situations, Pediatricians assume the role of Neonatal Resuscitation Program (NRP) providers and are responsible of the ETI procedure. They acquire this skill during residency training in the Neonatal Intensive Care Unit (NICU) and the delivery room. Difficulties in performing neonatal ETI lie in the small size of the mouth and airway of the neonate, and their particular anatomy of the larynx. This limited visibility represents a challenge even for the experienced clinician. Recently, a new videolaryngoscope (VL) technique has been introduced to the adult and pediatric medical fields as described respectively by Kaplan et al. and Weiss et al. In 2009, Vanderhal et al. reported a preliminary experience in the newborn population. Video assisted intubation could be a method of choice in teaching neonatal ETI.

To the best of our knowledge, there is no human study comparing the VL to the classic laryngoscope (CL) for acquiring the skill of neonatal ETI in the NICU.

This study aims:

1. To assess if the videolaryngoscope is superior to the classic laryngoscope in acquiring the neonatal endotracheal intubation skill in the Neonatal Intensive Care Unit; and
2. To assess if once the skill is acquired with the videolaryngoscope this experience is transferable to the use of the classic laryngoscope by showing a persistent difference in success rate in favor of the videolaryngoscope group.

The hypothesis are

1. Primary hypothesis:

   In the Neonatal Intensive Care Unit, use of the videolaryngoscope will increase success rate of endotracheal intubation by 20% compared to the classic laryngoscope. Later, acquired experience from the videolaryngoscope will be transferable to the use of the classic laryngoscope by showing a persistent difference in success rate of 20% in favor of the videolaryngoscope group.
2. Secondary hypothesis We expect that the videolaryngoscope will decrease time to intubation, and decrease rate of esophageal and right bronchial main stem intubations. It will also improve teaching of endotracheal intubations to pediatric residents by helping supervisors recognize problems related to intubation and by improving residents' level of confidence in performing the skill.

DETAILED DESCRIPTION:
Methodology

Consent to the study

The principal investigator will approach all pediatric residents to participate in the study. Parents of children will be approached by the principal investigator or the clinical research coordinator either antenatal or on admission to the NICU in the case of an eventual need for the infant of ETI. If the consent is made antenatally, we will insure that it is done by a different physician than the one performing the antenatal consultation.

Training to ETI

In our centre, residents learn neonatal ETI in the simulation centre at CHU Ste-Justine as first year residents when they are taught the NRP at the end of June every year, one week before starting residency training. The procedure is explained and demonstrated on a mannequin (Laerdal Neonatal Intubation Trainer) using the CL by a neonatologist and then residents practice on the same mannequin a couple of times (3-5). Further training is done in the clinical setting on real patients in an opportunistic manner. In both situations, they are supervised by a neonatologist or a senior subspecialty resident who will guide, coach and give them constructive feedback.

Residents who consent to the study will be trained to the use of the VL before randomization. This teaching session will be done similarly to the one described above. The procedure will be explained and demonstrated on a mannequin (Laerdal Neonatal Intubation Trainer) by the principal investigator using the VL and then residents will be offered to practice handling the VL and practice ETI on the same mannequin a couple of times (3-5). They will be supervised by the principal investigator who will guide, coach and give them constructive feedback. This process is to insure that residents depart with the same level of comfort (or discomfort) as the CL.

ETI procedure

In our unit, there are about two to three residents on service at a time. When a patient needs to be intubated priority goes to the resident who is in charge of that patient. In the case where the physician in charge is the neonatologist, the subspecialty resident or the nurse practitioner than a draw is done to decide which resident will proceed to the ETI. The pediatric resident is the first person to attempt an ETI and he is allowed three attempts. If he fails, the subspecialty resident, the respiratory therapist or the neonatologist proceed with the ETI. In the case of an urgent ETI (respiratory or cardiovascular instability, resuscitation, cardiovascular arrest, etc.) or complications during attempts by the resident, the senior physician (subspecialty resident or neonatologist) will proceed with the ETI.

At each ETI procedure, there is a resident, a neonatologist or a subspecialty resident, a nurse and a respiratory therapist. For the study, we will have a second respiratory therapist to assess our primary and secondary outcomes (using a stopwatch) and to collect the necessary data. About six respiratory therapists will be trained for this role, two per 8 hour shift. Monitoring of the child is done using a non invasive arterial blood pressure, an electrocardiogram and a pulse oximeter.

The devices used for the study will be the CL using Miller blades (size 0 and 1), and the C-MAC VL (blades size 0 and 1) developed by Karl Storz Endoscopy. The VL will be used to proceed to ETI indirectly with the use of the video monitor for guidance.

Premedication for ETI consists of a bolus of atropine 20 mcg/kg IV, fentanyl 2-5 mcg/kg diluted in 1 cc total of normal saline and given IV over 3 to 5 minutes, followed by a bolus of 2 mg/kg of IV succinylcholine. Facemask ventilation and preoxygenation is done before and between every attempt. After ETI, confirmation is done by auscultation and carbon dioxide detector, and a chest x-ray is performed to assess position of the tip of the endotracheal tube.

Definitions

1. Intubation is a success if the endotracheal tube is placed in the trachea under the vocal cords It is defined according to usual clinical norms: change in color of the carbon dioxide detector, vapor in the endotracheal tube, thoracic expansion, assessment of bilateral lung air entry, absence of air entry in the stomach by auscultation, and improvement of patient's clinical parameters: heart rate and arterial oxygen saturation.
2. Time to intubation is defined as the time from insertion of the laryngoscope blade in the patients' mouth until it is pulled out.
3. Esophageal intubation is diagnosed when there is absence of clinical signs of a successful endotracheal intubation and possibly air entry in the stomach by auscultation.
4. Right bronchial main stem intubation is diagnosed on chest x-ray.
5. A trial is counted as an attempt if there has been insertion of the laryngoscope blade in the patient's mouth.

Data collection for each intubation.

1. Patient: gestational age at birth, birth weight, sex of infant, post natal age, current weight, required inspired fraction of oxygen, number of ventilated days and number of previous intubations.
2. Intubator: training level, past training experience in pediatrics or neonatology, number of completed rotations in neonatology, and number of neonatal intubations tried, succeeded and failed in the past.
3. Intubation: date (later categorized into weekday and week-end), time (later categorized into day (8h-17h), evening (17h-00h) and night (00h-8h)), indication of intubation, semi urgent or elective intubation, number of attempts, length of each attempt, intubator for each attempt, final position of the tip of the endotracheal tube (including right bronchial main stem intubation), reason for failed intubation (including esophageal intubation), naso or orotracheal intubation, premedication used including doses and supervisor.
4. A survey will be distributed to the resident and the supervisor after each ETI event. The survey will assess the residents' level of confidence in attempting the ETI and will ask the supervisor the level of easiness in recognizing problems with laryngoscopy, endotracheal tube insertion and placement.

Randomization procedure

After consent, randomization will be done by distributing sealed envelopes and will be stratified according to the year of residency training. Residents will initially be randomized to intubate either with the videolaryngoscope (experimental group) or the classical laryngoscope (control group). In a second phase, all students will use the CL for ETI. Each resident is expected to perform at least five and a maximum of ten ETI per method. When a resident has reached ten ETI with the VL, he will change to the CL method. We are planning to obtain 100 ETI in each four groups for a total of 400 ETI.

Methods of data analysis and sample size estimates

Using the CL, the residents in our centre obtained a success rate of ETI of 55% (unpublished data). Assuming an increase of 20% of the success rate to 75% in the experimental group (VL), with an α level of 0.05 and a statistical power of 80%, we need 89 ETI per group. In the second phase, to show a 20% higher success rate in the experimental group (75%) than in the control group (55%) with the same statistical conditions, we need 89 more ETI per group for a total of 356 ETI. In the study, we plan to obtain 100 ETI per group for a total of 400 ETI. In our centre there are approximately 500 ETI a year. Of these, 20% (100) are done in the delivery room and another 20% (100) are done by the subspecialty resident, neonatologist or respiratory therapist because of urgency or difficulty of intubation. Considering a rate of patient recruitment of 60-75%, the study should be completed in 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Trainees: All residents registered in the three first years of the general pediatrics program of University of Montreal will be approached to participate in the study.
* Patients: All ETI attempted by pediatric residents in the NICU will be included in the study regardless of the patient weight or gestational age.

Exclusion Criteria:

* Trainees: Residents who perform less than five neonatal ETI per method.
* Patients: patients with major oral, cervical or upper airway malformations, urgent ETI with the inability to prepare in time the VL, and an unexpected difficult ETI.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation success rate. | 5 minutes

SECONDARY OUTCOMES:
Time to intubation. | 5 minutes
  Defined as the time from insertion of the laryngoscope blade in the patients' mouth until it is pulled out.
Rate of esophageal and right bronchial main stem intubations. | 15 minutes
  Esophageal intubation is diagnosed when there is absence of clinical signs of a successful endotracheal intubation and possibly air entry in the stomach by auscultation. Right bronchial main stem intubation is diagnosed on chest x-ray.
Supervisor's ease in recognizing problems with endotracheal intubation. | 15 minutes
  Short survey after each intubation.
Resident's level of confidence in attempting endotracheal intubation. | 15 minutes
  Short survey after each intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Moussa, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Dept Neonatology, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Moussa A, Luangxay Y, Tremblay S, Lavoie J, Aube G, Savoie E, Lachance C. Videolaryngoscope for Teaching Neonatal Endotracheal Intubation: A Randomized Controlled Trial. Pediatrics. 2016 Mar;137(3):e20152156. doi: 10.1542/peds.2015-2156. Epub 2016 Feb 12. PMID 26908701